CLINICAL TRIAL: NCT07266220
Title: Screening for Subclinical Atherosclerosis in Diabetic CKD Using Carotid Doppler
Brief Title: Carotid Doppler Screening for Subclinical Atherosclerosis in Diabetic CKD Patients.
Acronym: DiCKD-CAROTID
Status: Not yet recruiting | Type: Observational
Sponsor: Abdallah Ali Mohammed (Other)
Responsible Party: Sponsor-Investigator, Abdallah Ali Mohammed, Resident Physician, Internal Medicine, Assiut University
Organization: Assiut University (Other)
Other Study IDs: AUN-IM-CKD-CAROTID-2025
Record Dates: First submitted 2025-11-22; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 2; Chronic Kidney Disease; Atherosclerosis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is being done at Assiut University to look for early signs of hardening of the arteries (atherosclerosis) in people who have both diabetes and chronic kidney disease (CKD). Many patients with these conditions are at higher risk of heart disease and stroke, but the disease can develop quietly without symptoms.

We will use a safe, non-invasive test called carotid Doppler ultrasound, which uses sound waves to check the neck arteries (carotid arteries) for early changes. The goal is to see how often these early changes occur in patients with diabetes and CKD, and whether the findings relate to their kidney function, blood sugar control, and other health factors.

This research may help doctors detect vascular problems earlier and guide better prevention strategies for patients at risk.

ELIGIBILITY:
1. Age≥18years.
2. Diagnosis of type 2 diabetes mellitus (per treating physician or ADA criteria).
3. CKDstage3:eGFR30-59mL/min/1.73 m² on at least two measurements ≥3 months apart OR established diagnosis in medical record.
4. Clinically stable (no AKI, no hospitalization for cardiovascular event in past 3 months).
5. Ableandwilling to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with type 2 diabetes mellitus and stage 3 chronic kidney disease recruited from the nephrology and internal medicine outpatient clinics and inpatient wards of Assiut University Hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Prevalence of subclinical carotid atherosclerosis (defined as increased carotid intima-media thickness and/or carotid plaque detected by carotid Doppler ultrasound). | At baseline (single assessment at enrollment).
  Carotid Doppler ultrasound will be performed once at study entry to measure carotid intima-media thickness and detect the presence of carotid plaque. The percentage of patients with subclinical carotid atherosclerosis will be estimated among adults with type 2 diabetes mellitus and stage 3 chronic kidney disease.